CLINICAL TRIAL: NCT06262529
Title: Trajectories of Neurocognitive Impairment After Ischemic Stroke in Young Subjects
Brief Title: Neurocognitive Impairment After Ischemic Stroke
Acronym: COG-TRA-Y MRI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22-AOI-06
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Acute ischemic stroke (Experimental)
  Interventions: Other: Cerebral MRI

INTERVENTIONS:
Other: Cerebral MRI — Cerebral MRI at 72h / 3 months / 12 months

SUMMARY:
Affecting more than 150,000 patients in France, stroke is a major public health issue and a leading cause of disability worldwide. In western countries, 80-85% of strokes are of ischemic subtype. This study will focus on young adults, aged 18-45, with a diagnosis of ischemic stroke.

Studies assessing post-stroke cognition in young patients reported an alarming prevalence of cognitive impairment, affecting about 60% of stroke survivors between 4 and 12 months after the acute event. However, longitudinal data on neurocognitive trajectories (i.e., the evolution of cognitive impairment over time) in young patients with ischemic stroke are lacking. Collecting such data requires an exhaustive neuropsychological assessment and several functional evaluations, at different times, for the same patient.

Repeated neurocognitive study of young patients with ischemic stroke will enable: a description of the prevalence of impaired global cognitive efficiency, an analysis of the specific neurocognitive domains affected, and the tracing of trajectories of recovery from cognitive impairment over time, in terms of global cognitive efficiency and as a function of specific neurocognitive domains (memory, executive, attentional, social cognition, instrumental functions, fatigability, etc.).

Up to date, the clinic-radiological predictors and associated factors of neurocognitive impairment after ischemic stroke in young patients have not been studied. Ischemic stroke causes acute brain lesions of the gray matter (GM) and white matter (WM). Numerous studies suggest that cognitive health may be more closely linked to the integrity of WM than to GM. Magnetic resonance imaging (MRI), and in particular diffusion tensor imaging (DTI) sequences, analyze WM bundles. By using fiber tracking algorithms image analysis enable the WM fiber bundle reconstruction and allow quantifying the volume of lesions (pre-existing and ischemic stroke-induced) in the WM tract.

The aim of this study is to study whether the extension of pre-existing and acute white matter lesions is associated with poorer cognitive recovery after ischemic stroke, both in terms of global cognitive performance and impairment in specific neurocognitive domains.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 45 years.
* Pathology: ischemic stroke diagnosed with brain MRI as per standard clinical practice, with or without occlusion of proximal artery, anterior or posterior circulation.
* Ability to understand and complete study tests and questionnaires: fluent French speaker and reader.
* All patients must be affiliated to a social security scheme.
* Signature of informed consent form.

Exclusion Criteria:

* Pre-existing cognitive impairment (defined as CQI <78 or clinical dementia).
* Severe functional dependence prior to stroke (defined as Modified Rankin Scale MRS = score 5).
* Any neurological or psychiatric comorbidity.
* Sensory disorders: visual impairment, blindness, deafness.
* Severe acquired phasic disorders: on the expressive oral side, in the presence of an inability to express oneself, which interferes with the collection of responses to neuropsychological tests; and on the receptive oral side, in the presence of an inability to understand the instructions of neuropsychological tests. Phasic functioning is systematically assessed during hospitalization by means of the NIHSS (score ≤ 2 on the "Language" sub-test), and will be rechecked clinically and psychometrically during neuropsychological assessments using the Language Screening Test (LAST) for both expression and oral comprehension. - Severe motor disorders: inability to mobilize the dominant upper limb for written neuropsychological tests.
* Contraindication to MRI.
* Pregnant women.
* HIV-positive patients: interaction of infectious pathology on cognitive functioning. Declarative, no HIV tests will be performed.
* Withdrawal of informed consent.
* Consumption of alcohol and/or narcotics on the day of neuropsychological assessments.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2025-05-09 (Estimated); Study Completion 2027-05-09 (Estimated)

PRIMARY OUTCOMES:
evolution of neurocognitive disorders (trajectories of global cognitive efficiency) over 1 year after stroke | Between 3 months and 12 months
  Montréal cognitive assessment (MOCA - score 0 to 30)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - cannes Hospital, Cannes
  - Nice University Hospital, Nice

IPD SHARING:
Plan to Share IPD: No